CLINICAL TRIAL: NCT00511992
Title: Phase II Study of Paclitaxel (TAXOL), Intraperitoneal Cisplatin and IV Avastin Followed by Avastin Consolidation for Advanced Ovarian and Peritoneal Carcinoma or Fallopian Tube Cancer
Brief Title: Study of Bevacizumab Followed by Bevacizumab Consolidation for Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2674
Record Dates: First submitted 2007-08-03; First posted 2007-08-06 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Advanced Ovarian Carcinoma; Primary Peritoneal Carcinoma; Ovarian Carcinosarcoma
Keywords: Ovarian Cancer; Gynecologic Cancer; Ovarian Carcinoma; Peritoneal Carcinoma; IP chemotherapy; Intraperitoneal; Avastin; Bevacizumab
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Bevacizumab; Paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Avastin (Experimental)
  Interventions: Drug: Avastin; Drug: Paclitaxel; Drug: Cisplatin

INTERVENTIONS:
Drug: Avastin — Initial Treatment Bevacizumab 15mg/kg Day 1 IV every 21 days x 5 cycles (beginning with cycle 2)
  Consolidation Treatment:
  Avastin 15mg/kg IV every 21 days x 12 cycles
  Other Names: Bevacizumab
Drug: Paclitaxel — Paclitaxel 135mg/m2 IV Day 1 every 21 days x 6 cycles
Drug: Cisplatin — 75mg/m2 IP day 2 every 21 days x 6 cycles

SUMMARY:
The purpose of this study is to evaluate the tolerability of intraperitoneal cisplatin with intravenous paclitaxel and Avastin as defined by the proportion of patients able to complete 6 cycles of treatment.

DETAILED DESCRIPTION:
Ovarian cancer is the leading cause of death from gynecologic cancer in the United States. The high death rate stems from late presentation and tumor that has spread beyond the ovary at the time of diagnoses.

Ovarian cancer typically spreads throughout the peritoneal cavity. Three randomized clinical trial have recently demonstrated the superiority of intraperitoneal(IP) over intravenous platinum based chemotherapy in optimally debulked advance ovarian cancer. The success of Bevacizumab in metastatic colorectal cancer has led to trials evaluating its' efficacy in advanced ovarian cancer. Based on the mechanism of action of Bevacizumab, there may be benefit of extended therapy with this agent.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage II and III epithelial ovarian carcinoma, primary peritoneal carcinoma, or ovarian carcinosarcoma.
* Adequate bone marrow, renal, and hepatic function
* Patients must be entered no more than twelve weeks postoperatively

Exclusion Criteria:

* Patients with epithelial ovarian carcinoma of low malignant potential (borderline carcinomas).
* Stage IV or suboptimally debulked disease following primary cytoreductive surgery
* Patients who have received prior radiotherapy or chemotherapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-07; Primary Completion 2015-08-03 (Actual); Study Completion 2015-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: D. Scott McMeekin, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Avastin: Avastin: Initial Treatment:
  Paclitaxel 135mg/m2 IV Day 1 every 21 days x 6 cycles, Cisplatin 75mg/m2 IP Day 2 every 21 days x 6 cycles, Bevacizumab 15mg/kg Day 1 IV every 21 days x 5 cycles (beginning with cycle 2)
  Consolidation Treatment:
  Avastin 15mg/kg IV every 21 days x 12 cycles
Period: Overall Study
Arm/Group | Avastin
Started | 20
Completed | 13
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Avastin
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 6
Age, Continuous [Mean (Full Range); unit: years] | 59 [45 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Able to Complete 6 Cycles of Treatment.
Description: Completion of cycle 6
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Avastin
Number analyzed (Participants) | 20
Participants | 17

2. Secondary Outcome: Number of Patients Who Experienced Toxicities Associated With Intraperitoneal Cisplatin With Intravenous Paclitaxel and Avastin.
Description: CTCAE assessment of toxicity
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Avastin
Number analyzed (Participants) | 20
Participants | 2

ADVERSE EVENTS:
Time Frame: 6 years
Arm/Group | Avastin
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 2/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avastin (N=20)
Entero-vesical fistula (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avastin (N=20)
Grade 3 Neurpoathy (Nervous system disorders) | 1 (1)
Grade 3 abdominal pain (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes